CLINICAL TRIAL: NCT01851642
Title: The Role of Conformational Diseases on Macrophage Function
Brief Title: Lung Disease and Its Affect on the Work of White Blood Cells in the Lungs
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201501051; 699 (Other: Shands UF Clinical Research Center); 08-2007 (Other: University of Florida)
Record Dates: First submitted 2013-04-25; First posted 2013-05-10 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Alpha-1 Antitrypsin Deficiency; AAT Deficiency; AATD; Cystic Fibrosis (CF)
Keywords: Macrophage; Alpha-1 Antitrypsin Deficiency; Cystic Fibrosis
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Cystic Fibrosis | interventions — Health Records, Personal; Restraint, Physical; Blood Specimen Collection; Phlebotomy; Respiratory Physiological Phenomena; Albuterol; Procaterol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AAT Deficiency: Those diagnosed with Alpha-1 Antitrypsin (AAT) Deficiency. At every study visit, a history and physical exam (H&P), blood draw, and pulmonary function testing (PFTs) with the use of an albuterol inhaler will be done.
  Interventions: Procedure: History and physical exam.; Procedure: Blood draw.; Procedure: Pulmonary function testing.; Drug: Albuterol inhaler.
- Cystic Fibrosis: Those diagnosed with Cystic Fibrosis (CF) with mutation Delta F508. At every study visit, a history and physical exam (H&P), blood draw, and pulmonary function testing (PFTs) with the use of an albuterol inhaler will be done.
  Interventions: Procedure: History and physical exam.; Procedure: Blood draw.; Procedure: Pulmonary function testing.; Drug: Albuterol inhaler.
- Without Lung Disease Diagnosis: Those without the diagnosis of AAT Deficiency or CF. At every study visit, a history and physical exam (H&P), blood draw, and pulmonary function testing (PFTs) with the use of an albuterol inhaler will be done.
  Interventions: Procedure: History and physical exam.; Procedure: Blood draw.; Procedure: Pulmonary function testing.; Drug: Albuterol inhaler.

INTERVENTIONS:
Procedure: History and physical exam. — At every study visit, participant's will be asked about their medical history and will have a physical exam.
  Other Names: H&P
Procedure: Blood draw. — At each study visit, participants will have an intravenous catheter (IV) placed in one of their veins and blood will be drawn from the IV for study testing.
  Other Names: Phlebotomy
Procedure: Pulmonary function testing. — At every study visit, participants will have their lung function assessed. This is done by blowing forcefully at least 3 times into a tube. Testing will be done two times; before and after the use of an Albuterol inhaler.
  Other Names: PFTs
Drug: Albuterol inhaler. — At every study visit, participating subjects will take 2 puffs of an Albuterol inhaler after the first set of PFTs, but before the second set of PFTs. There will be at least a 30 minute period after the use of the Albuterol inhaler and the second set of PFTs.
  Other Names: Ventolin; Proventil; Proventil-HFA; AccuNeb; Vospire; ProAir

SUMMARY:
The purpose of this study is to look at how Alpha-1-antitrypsin (AAT) deficiency and Cystic Fibrosis (CF) affect white blood cells in the lungs, called macrophages, and their ability to work.

DETAILED DESCRIPTION:
AAT deficiency is a genetic disorder that affects around 100,000 people in the USA, including 1-3% of all people diagnosed with chronic obstructive pulmonary disease (COPD). In AAT deficient people diagnosed with COPD, it was originally believed the cause of the disease was due to a lack of supply of alpha-1 antitrypsin. However, early information gathered in our laboratory suggests another cause of the development of COPD and the progressing of the disease may be due to a malfunction in macrophages.

CF is also a genetic disorder which affects 1/300 births among the Caucasian population. One of the main symptoms of CF is inflammation of the lung tissue. Lung macrophages play a major role in lung inflammation as well as in helping to resolve the inflammation.

Inflammation is an important defense of the body. It is the body's response to infection causing germs and things that may cause irritation, as well as, a way for the body to repair damaged tissue.

We suggest that the effects of AAT deficiency and CF decreases the inflammation response in the lungs and also restricts the ability of macrophages to correct that inflammation once it occurs.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female 18 years of age or older
* Negative pregnancy test for women of childbearing potential
* Hemoglobin >12.5 g/dl measured on the day of participation
* Negative urine nicotine test

Exclusion Criteria:

* Pregnancy or breastfeeding
* Weight < 50 kg
* History of anemia requiring blood transfusions, erythropoietin supplementation, or iron supplementation within the past 36 months
* Known hemoglobin <12.5 g/dl within the past 90 days
* Systolic blood pressure > 180 mmHg and/or diastolic blood pressure >100 mmHg
* Poor venous access
* Large volume blood donation (>200 ml or 7 ounces) within the previous 56 days (e.g. blood donation for the purposes of blood banking)
* Clinically significant cardiac, hemostatic or neurological impairment or any other significant medical condition that, in the opinion of the investigator would affect subject safety (e.g., recent myocardial infarction, history of prolonged bleeding time, cerebral vascular accident, advanced cancer or uncontrolled medical condition)
* Psychiatric or cognitive disturbance or illness that would affect subject safety
* Current smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Alpha-1 Antitrypsin (AAT) Deficient subjects, Cystic Fibrosis(CF) subjects with mutation Delta F508, and subjects without either diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2007-08-09 (Actual); Primary Completion 2032-07-20 (Estimated); Study Completion 2033-07-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of macrophage function. | On average, within 30 days from the time the blood is collected.
  From every study participant, we will collect blood from a vein through the placement of an intravenous catheter (IV). We will complete various experiments that will allow us to see how well each participant's macrophage cells are working.

SECONDARY OUTCOMES:
Comparison of the amount of alpha-1 antitrypsin in the blood. | On average, within 30 days from the time the blood was collected.
  From every study participant, we will collect blood from a vein through an IV.
Comparison of the amount of an inflammatory marker in the blood, called C-reactive protein. | On average, within 30 days from the time the blood is collected.
  From every study participant, we will collect blood from a vein through and IV.
Evaluation of lung function. | On average, within 30 days from the time the testing is completed.
  Lung function testing will be done on every study participant. This is is done by forcefully blowing into a tube on at least 3 separate occasions. Albuterol, an inhaled medication used to expand lung airways, will be given after lung function testing and then the testing will be repeated after 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Karina Serban, MD, Principal Investigator — University of Florida, College of Medicine, Division of Pulmonary, Critical Care, and Sleep Medicine
Locations (1):
- Shands at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Enrolled subjects may request a copy of their clinical testing done while enrolled in the clinical trial. All other data used for publication purposes will be de-identified.
Time Frame: This study is a tissue data bank study and data will not be shared with the public
Access Criteria: This is no sharing of data in this tissue banking study, so no share access will be used

REFERENCES:
- [Background] Blank CA, Brantly M. Clinical features and molecular characteristics of alpha 1-antitrypsin deficiency. Ann Allergy. 1994 Feb;72(2):105-20; quiz 120-2. PMID 8109800
- [Background] Yoshida A, Lieberman J, Gaidulis L, Ewing C. Molecular abnormality of human alpha1-antitrypsin variant (Pi-ZZ) associated with plasma activity deficiency. Proc Natl Acad Sci U S A. 1976 Apr;73(4):1324-8. doi: 10.1073/pnas.73.4.1324. PMID 1083527
- [Background] Jeppsson JO. Amino acid substitution Glu leads to Lys alpha1-antitrypsin PiZ. FEBS Lett. 1976 Jun 1;65(2):195-7. doi: 10.1016/0014-5793(76)80478-4. No abstract available. PMID 1084290
- [Background] Lomas DA, Evans DL, Finch JT, Carrell RW. The mechanism of Z alpha 1-antitrypsin accumulation in the liver. Nature. 1992 Jun 18;357(6379):605-7. doi: 10.1038/357605a0. PMID 1608473
- [Background] Perlmutter DH. Liver injury in alpha1-antitrypsin deficiency: an aggregated protein induces mitochondrial injury. J Clin Invest. 2002 Dec;110(11):1579-83. doi: 10.1172/JCI16787. No abstract available. PMID 12464659
- [Background] Hidvegi T, Schmidt BZ, Hale P, Perlmutter DH. Accumulation of mutant alpha1-antitrypsin Z in the endoplasmic reticulum activates caspases-4 and -12, NFkappaB, and BAP31 but not the unfolded protein response. J Biol Chem. 2005 Nov 25;280(47):39002-15. doi: 10.1074/jbc.M508652200. Epub 2005 Sep 23. PMID 16183649
- [Background] Kaufman RJ. Orchestrating the unfolded protein response in health and disease. J Clin Invest. 2002 Nov;110(10):1389-98. doi: 10.1172/JCI16886. No abstract available. PMID 12438434
- [Background] Oda Y, Okada T, Yoshida H, Kaufman RJ, Nagata K, Mori K. Derlin-2 and Derlin-3 are regulated by the mammalian unfolded protein response and are required for ER-associated degradation. J Cell Biol. 2006 Jan 30;172(3):383-93. doi: 10.1083/jcb.200507057. PMID 16449189
- [Background] Seager Danciger J, Lutz M, Hama S, Cruz D, Castrillo A, Lazaro J, Phillips R, Premack B, Berliner J. Method for large scale isolation, culture and cryopreservation of human monocytes suitable for chemotaxis, cellular adhesion assays, macrophage and dendritic cell differentiation. J Immunol Methods. 2004 May;288(1-2):123-34. doi: 10.1016/j.jim.2004.03.003. PMID 15183091
- [Background] Newman BH. Donor reactions and injuries from whole blood donation. Transfus Med Rev. 1997 Jan;11(1):64-75. doi: 10.1016/s0887-7963(97)80011-9. PMID 9031492
- See also: University of Florida, Division of Pulmonary Medicine, Critical Care & Sleep Medicine — http://pulmonary.medicine.ufl.edu/